CLINICAL TRIAL: NCT06923657
Title: Application of PSMA PET/MRI-guided Prostate Targeted Biopsy in Patients With PI-RADS ≤ 3 and Negative Previous Biopsy: A Single-center, Prospective, Open-label, Randomized Controlled Trial
Brief Title: PSMA PET/MRI-Guided Prostate Biopsy for PI-RADS ≤3 and Prior Negative Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ning Xu, Deputy Director of Department, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MRCTA,ECFAH OfFMU[2024]837
Record Dates: First submitted 2025-03-26; First posted 2025-04-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer Screening; PSMA-PET
Keywords: imaging examinations; PSMA PET/MRI; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The control group (Active Comparator): The control group will receive TRUS guided transperineal saturation biopsy.
  Interventions: Diagnostic Test: TRUS guided transperineal saturation biopsy
- The experimental group (Experimental): The experimental group will undergo PSMA PET/MRI examination. For those with positive PSMA PET/MRI results, a PSMA PET/MRI-TRUS guided prostate targeted biopsy will be performed based on transrectal ultrasound (TRUS) guided transperineal saturation biopsy, targeting the positive lesions. For those with negative PSMA PET/MRI results, only TRUS guided transperineal saturation biopsy will be performed.
  Interventions: Diagnostic Test: PSMA PET/MRI-TRUS guided prostate targeted combined saturation biopsy

INTERVENTIONS:
Diagnostic Test: PSMA PET/MRI-TRUS guided prostate targeted combined saturation biopsy — The experimental group will undergo PSMA PET/MRI examination. For those with positive PSMA PET/MRI results, a PSMA PET/MRI-TRUS guided prostate targeted biopsy will be performed based on transrectal ultrasound (TRUS) guided transperineal saturation biopsy, targeting the positive lesions. For those with negative PSMA PET/MRI results, only TRUS guided transperineal saturation biopsy will be performed. Clinical and pathological data of the patients will be collected for statistical analysis.
  Arms: The experimental group
Diagnostic Test: TRUS guided transperineal saturation biopsy — The control group will receive TRUS guided transperineal saturation biopsy. Clinical and pathological data of the patients will be collected for statistical analysis.
  Arms: The control group

SUMMARY:
The goal is to provide more accurate diagnostic tools and optimized diagnostic workflows for clinically suspected prostate cancer patients with prior negative biopsies, improving early detection rates for csPCa and reducing missed diagnoses.

DETAILED DESCRIPTION:
This research intends to prospectively enroll patients with prior negative biopsies, a PI-RADS score ≤ 3, and persistent PSA or PHI elevation, randomly assigning them to the PSMA PET/MRI group (experimental group) and the TRUS-guided transperineal saturation biopsy group (control group). The research aims to evaluate the application of PSMA PET/MRI in clinically suspected prostate cancer patients with prior negative biopsies, comparing the differences in csPCa detection rates between PSMA PET/MRI-TRUS guided prostate targeted biopsy and TRUS-guided saturation biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Serum PSA > 4 ng/mL
* At least one prior negative prostate biopsy
* At least two consecutive increases in PSA and/or PHI
* Negative digital rectal examination
* Multiparametric MRI (mpMRI) indicating a PI-RADS score ≤ 3

Exclusion Criteria

* Age ≤ 30 years or > 85 years
* Concurrent presence of other malignant tumors
* Previous treatment with any form of anti-tumor therapy or prostate surgery (excluding prostate biopsy)
* Inability to comply with PSMA PET/MRI examination (e.g., contrast allergy, claustrophobia, etc.)
* Contraindications for prostate biopsy (e.g., coagulation disorders, acute prostatitis, acute urinary tract infection, etc.)
* Severe organ dysfunction (e.g., significant cardiac, pulmonary, hepatic, or renal impairment)
* Incomplete clinical or pathological data

Ages: 30 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Sensitivity | Perioperative
  It refers to the percentage of patients who actually have prostate cancer correctly identified as positive (true positive). The calculation formula is: TP/(TP+FN)×100%. TP is true positive, and FN is false negative.
Diagnostic Specificity | Perioperative
  It refers to the percentage of patients who do not actually have prostate cancer correctly identified as negative (true negative). The calculation formula is: TN/(TN+FP)×100%. TN is true negative, and FP is false positive.
Positive Predictive Value(PPV) | Perioperative
  It refers to the proportion of true positives among the positive results obtained by a specific testing method. The calculation formula is: PPV = TP/(TP+FP)×100%.
Negative Predictive Value(NPV) | Perioperative
  It refers to the proportion of true negatives among the negative results obtained by a specific testing method. The calculation formula is: NPV = TN/(TN+FN)×100%.
Positive Likelihood Ratio(PLR) | Perioperative
  It refers to the ratio of the probability of correctly identifying a patient with prostate cancer as positive to the probability of incorrectly identifying a patient without prostate cancer as positive. The calculation formula is: +LR = Sensitivity / (1- Specificity)×100%.
Negative Likelihood Ratio(NLR) | Perioperative
  It refers to the ratio of the probability of incorrectly identifying a patient with prostate cancer as negative to the probability of correctly identifying a patient without prostate cancer as negative. The calculation formula is:-LR = (1- Sensitivity) / Specificity×100%.
Correct Diagnostic Index | Perioperative
  It refers to the sum of sensitivity and specificity minus 1. The correct diagnostic index can be used for comparing two diagnostic methods, with an ideal correct diagnostic index of 100%.r = (Specificity+Sensitivity) -1 = 1- (False Positive Rate + False Negative Rate).

SECONDARY OUTCOMES:
PRECISION Questionnaire | 1 week before biopsy, 1 week after biopsy, 1 month, 3 months, 6 months, 12 months.
  The incidence of complications for the two biopsy methods.
EORTC QLQ-C30 Questionnaire | Before diagnosis, 1 month, 3 months, 6 months, 12 months
  The change in quality of life compared to baseline values in the experimental group and control group.
Generalized Anxiety Disorder GAD-7 Scale | Before diagnosis, 1 week after diagnosis, 1 month, 3 months, 6 months, 12 months
  The difference in anxiety levels at each time point between the experimental group and the control group.
Decision Conflict Scale, Decision Regret Scale | Before diagnosis, 1 month, 3 months, 6 months
  The decision-making differences at each time point between the experimental group and the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No